CLINICAL TRIAL: NCT00171938
Title: Open-label Trial of Imatinib Mesylate in Patients With Unresectable Recurrent Glioblastoma Multiforme Expressing PDGFR (Platelet Derived Growth Factor Receptors)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BBR03
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2009-11

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Brain tumors; Imatinib; PDGFR
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
This is an open label clinical trial of imatinib mesylate 800 mg po/day in a population of patients with unresectable, recurrent glioblastoma multiforme. Patients will be treated for up to 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented diagnosis of GBM.
2. Immunohistochemical documentation of expression of PDGFR.
3. Unresectable, recurrent disease by MRI and spectroscopy

Exclusion Criteria:

1. Treatment with any other investigational agents within 28 days of first day of study drug dosing.
2. Concurrent chemotherapy.
3. Concurrent radiotherapy.

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
PFS (progression free-survival), defined by the percentage of patients without evidence of progressive disease in 6 months

SECONDARY OUTCOMES:
Objective Tumoral Response defined by RECISt criteria performed by MRI
OS (overall survival)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Rio Grande, Brazil